CLINICAL TRIAL: NCT04896775
Title: NiteCAPP: Web-based Interventions for Insomnia in Rural Dementia Caregivers: Examination of Sleep, Arousal, Mood, Cognitive, and Immune Outcomes
Brief Title: NiteCAPP: Web-based Interventions for Insomnia in Rural Dementia Caregivers
Acronym: NiteCAPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY004494
Record Dates: First submitted 2021-05-05; First posted 2021-05-21 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Insomnia; Dementia
Keywords: Dementia Caregiver
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NiteCAPP CARES (Experimental): Cognitive Behavioral Treatment-Insomnia. Web-based intervention that will include 4 weekly sessions and 4 bimonthly boosters. Each session is to be completed individually by CG (with PWD to extent able) in a single sitting (less than 45 mins). Each session should be completed in 7 days with next session released only after prior one completed. Session 1 focuses on sleep education, sleep hygiene, and stimulus control. Session 2 focuses on sleep compression, relaxation, and problem solving. Session 3 focuses on coping and stress management and cognitive therapy. Session 4 focuses on a review of skills and plan for maintenance of behavior change.
  Interventions: Behavioral: NiteCAPP CARES
- NiteCAPP SHARES (Experimental): Sleep Hygiene and Related Education. Web-based intervention that will include 4 weekly sessions and 4 bimonthly boosters. Each session is to be completed individually by CG (with PWD to extent able) in a single sitting (less than 45 mins). Each session should be completed in 7 days with next session released only after prior one completed. Session 1 focuses on expanded sleep education and sleep hygiene. Session 2 focuses insomnia education and sleep hygiene support. Session 3 focuses on targeted sleep education and sleep in dementia. Session 4 focuses on a review of skills and plan for maintenance of behavior change. Boosters review skills, encourage practice, and troubleshoot issues.
  Interventions: Behavioral: NiteCAPP SHARES

INTERVENTIONS:
Behavioral: NiteCAPP CARES — Web-based intervention that will include 4 weekly sessions and 4 bimonthly boosters. Each session is to be completed individually by CG (with PWD to extent able) in a single sitting (less than 45 mins). Each session should be completed in 7 days with next session released only after prior one completed. Session 1 focuses on sleep education, sleep hygiene, and stimulus control. Session 2 focuses on sleep compression, relaxation, and problem solving. Session 3 focuses on coping and stress management and cognitive therapy. Session 4 focuses on a review of skills and plan for maintenance of behavior change.
  Other Names: Web CBT-I
  Arms: NiteCAPP CARES
Behavioral: NiteCAPP SHARES — Web-based intervention that will include 4 weekly sessions and 4 bimonthly boosters. Each session is to be completed individually by CG (with PWD to extent able) in a single sitting (less than 45 mins). Each session should be completed in 7 days with next session released only after prior one completed. Session 1 focuses on expanded sleep education and sleep hygiene. Session 2 focuses insomnia education and sleep hygiene support. Session 3 focuses on targeted sleep education and sleep in dementia. Session 4 focuses on a review of skills and plan for maintenance of behavior change. Boosters review skills, encourage practice, and troubleshoot issues.
  Other Names: Web Sleep Hygiene and Related Education (Web-SHARE)
  Arms: NiteCAPP SHARES

SUMMARY:
The goal of this project evaluate the efficacy of NiteCAPP in improving insomnia in a rural dementia caregiver sample (n of 100 caregiver and PWD dyads). We will measure both the short term (post-treatment) and long term (6 and 12 months) effects of the intervention on CG sleep, arousal, inflammation, health, mood, burden and cognitive function, and PWD sleep.

DETAILED DESCRIPTION:
Over the next 30 years, more than 10 million persons living with dementia in the US will receive care at home from an unpaid and untrained family caregiver. At home care is preferred by caregivers (CG) and persons with dementia (PWD) alike, but increases caregiver risk of insomnia and related negative health outcomes, including depression, anxiety, cognitive disturbances and poor quality of life. Cognitive behavioral therapy for insomnia (CBT-I) is an effective and established evidence based treatment for adults of all ages. Although relatively understudied in dementia caregivers, the research suggests CBT-I is also efficacious in caregivers. Our team developed a brief (4 session) CBT-I protocol adapted for dementia caregivers and has shown in person and remote (i.e. telehealth) delivery of this protocol significantly reduces insomnia and improves mood (moderate to large effects). Given demands on caregiver time and limited availability of trained CBT-I providers, we developed a web-based version of this treatment (NiteCAPP) to increase accessibility of this efficacious treatment for rural dementia CGs. NiteCAPP will allow for flexible at home scheduling, and the skills needed to monitor caregiver treatment progress can be quickly and efficiently taught to healthcare providers. The Cognitive Activation Theory of Stress provides a framework for our basic premise that CGs experience insomnia, arousal and inflammation that prompt sympathetic activation and hypothalamic-pituitary-adrenal (HPA) disruption that have negative effects on health. The proposed trial tests the novel hypothesis that NiteCAPP will improve CG health, mood, burden and cognition by targeting their shared mechanisms - sleep, arousal and inflammation - thereby, returning sympathetic and HPA functioning to normal. Another novel aspect of the proposed trial is inclusion of behavioral strategies to target the PWD sleep. Objectives: The goal of this project evaluate the efficacy of NiteCAPP in improving insomnia in a rural dementia caregiver sample (n of 100 caregiver and PWD dyads). We will measure both the short term (post-treatment) and long term (6 and 12 months) effects of the intervention on CG sleep, arousal, inflammation, health, mood, burden and cognitive function, and PWD sleep.

ELIGIBILITY:
Inclusion:

Caregiver Eligibility. Inclusion criteria: 1. 18+ yrs, 2. CG living with PWD, 3. willing to be randomized, 4. read/understand English, 5. insomnia diagnosis, 6. no prescribed or over the counter sleep meds for 1+ mo, or stabilized 6+ mos.

* Insomnia: 1. complaints for 6+ mos, 2. adequate opportunity and circumstances for sleep, 3. 1+ of the following: difficulty falling asleep, staying asleep or waking too early, 4. daytime dysfunction (mood, cognitive, social, occupational) due to insomnia, 5. baseline diaries indicate >30 mins of sleep onset latency or wake after sleep onset on 3+ nts.

PWD Eligibility. 1. probable/possible Alzheimer's Disease (self-report or primary care provider written confirm), 2. 1+ problem on Nighttime Behavior Inv. 3+ nts/wk, 3. tolerate actigraphy, 4. no sleep meds 1+ mo or stabilized 6+ mos, 5. untreated sleep disorder for which CBT-I is not recommended (e.g., apnea), 6. scoring <32 on Sleep Apnea scale, Sleep Disorders Ques.

Exclusion:

CG Exclusion criteria: 1. unable to consent, 2. cognitive impairment [Telephone Interview for Cognitive Status (TICS) <25], 3. sleep disorder other than insomnia [i.e., apnea (apnea/hypopnea index-AHI >15)], 4. bipolar or seizure disorder, 5. other major psychopathology except depression or anxiety (e.g., suicidal, psychotic), 6. severe untreated psychiatric comorbidity, 7. psychotropic or other medications (e.g., beta-blockers) that alter sleep, 8. non-pharmacological tx for sleep or mood outside current trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-02-02 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Completion | Single administration at 8 weeks
  Percentage of sessions completed out of the 4 sessions/modules included in NiteCAPP and WebSHE.
Adherence | Single administration at 8 weeks
  Percentage of the intervention instructions followed as indicated on the treatment adherence logs completed each day during treatment.
Internet Intervention Utility Questionnaire | Single administration at 8 weeks
  Questionnaire with 15 items, including two open-ended questions, that assesses the usability, like-ability, and usefulness of online interventions using a 5-point Likert scale from 1-not at all to 5-very. The two open-ended questions ask the participant to list the most and least helpful parts of the program
Satisfaction Survey | Single administration at 8 weeks
  Survey that assesses the patient's experience and satisfaction with treatment.
Insomnia Severity Index | Single administration at baseline, 8 weeks, 6 month and 12 follow up
  Brief self-report measure of current perception of insomnia symptom severity, distress and daytime impairment. Commonly used as an outcome assessment in insomnia treatment research.
Daily Electronic Sleep Diaries | Daily at baseline, 8 weeks, 6 month and 12 follow up
  Completed each morning (~5 mins) during each assessment period. Electronic daily diaries collecting self-reported information on caregiver sleep onset latency (time to fall asleep), wake after sleep onset (time awake after sleep onset to last awakening), and sleep efficiency (total sleep time divided by time in bed and multiplied by 100). We developed and tested these electronic diaries.
Change in Pain Intensity - Daily Electronic Sleep Diaries | Daily at baseline, 8 weeks, 6 month and 12 follow up
  Daily electronic dairies will record pain intensity; range: 0-100 (no pain- most intense)
Change in Pain Unpleasantness - Daily Electronic Sleep Diaries | Daily at baseline, 8 weeks, 6 month and 12 follow up
  Daily electronic dairies will record pain unpleasantness; range: 0-100 (none- most unpleasantness)
Change in Wake After Sleep Onset - Daily Electronic Sleep Diaries | Daily at baseline, 8 weeks, 6 month and 12 follow up
  Daily electronic dairies will record wake after sleep onset (number of minutes)
Change in Sleep Onset Latency- Daily Electronic Sleep Diaries | Daily at baseline, 8 weeks, 6 month and 12 follow up
  Daily electronic dairies will record sleep onset latency (number of minutes)
Change in Sleep Efficiency- Daily Electronic Sleep Diaries | Daily at baseline, 8 weeks, 6 month and 12 follow up
  Daily electronic dairies will record sleep efficiency
Change in Fatigue - Daily Electronic Sleep Diaries | Daily at baseline, 8 weeks, 6 month and 12 follow up
  Daily electronic dairies will record insomnia severity; range: 0-100 (no insomnia - most severe)
Change in Sleep and Pain Medication - Daily Electronic Sleep Diaries | Daily at baseline, 8 weeks, 6 month and 12 follow up
  Daily electronic dairies will record daily medication consumption
Change in Perceived Stress Scale | Single administration at baseline, 8 weeks, 6 month and 12 follow up
  Perceived Stress Scale is a self-report measure of how life situations are perceived as stressful. The scale consists of 15 items corresponding to everyday situation and participants are asked to rate on a Likert scale from 0 (never) to 4 (very often) how
Change in Kingston Caregiver Stress Scale (KCSS) | Single administration at baseline, 8 weeks, 6 month and 12 follow up
  A 10-item scale that asks caregivers to rate on a scale from 1 (no stress) to 5 (extreme stress) how much stress they experience related to various aspects of caregiving.
Change in Dysfunctional Beliefs About Sleep (DBAS) | Single administration at baseline, 8 weeks, 6 month and 12 follow up
  A self-report measure of sleep-related arousal. This measure consists of 30 questions intended to measure 5 dimensions: misconceptions about the causes of insomnia, misattributions or amplifications of the consequences, unrealistic expectations, control, and predictability of sleep and faulty beliefs about sleep promoting practices. Although the original scale used a 100 mm VAS, subsequent research with the DBAS has used an 11-point Likert scale (0 = strongly disagree, 10 = strongly agree), and the latter response method will be used.
Change in Peripheral Arousal | Single administration at baseline, 8 weeks, 6 month and 12 follow up
  Holter monitor assessed 5 min ECG recordings at rest at home (enhancing ecological validity). Variables: RMSDNN (root mean sqrd standard dev. of N-N intervals), pNN50 (percent of N-N intervals less than 50 ms), LF over HF (high frequency divided by low frequency ratio; index of autonomic nervous system regulation).
Change in Inflammation | Single blood draw at baseline, 8 weeks, 6 month and 12 follow up
  Blood based biomarkers will be examined at each assessment period. Biomarkers include: inflammatory (HS-CRP, IL-6), neurodegenerative ( AβB42, tau levels)
Change in Blood-based Biomarker Interleukin 6 IL-6) | Single blood draw at baseline, 8 weeks, 6 month and 12 follow up
  Inflammation
Change in Blood-based Biomarker AβB42 | Single blood draw at baseline, 8 weeks, 6 month and 12 follow up
  Neurodegenerative
Change in Blood-based Biomarker Tau | Single blood draw at baseline, 8 weeks, 6 month and 12 follow up
  Neurodegenerative

SECONDARY OUTCOMES:
Change in State-Trait Anxiety Inventory (STAI) | Single administration at baseline, 8 weeks, 6 month and 12 follow up
  Inventory that asks respondents to rate how true 20 self-descriptive statements (e.g., I feel calm) are on a 4-point scale (1 = not at all, 4 = very much so). Typically, respondents are asked to rate statements according to how they generally feel (trait-anxiety scale) and how they feel in the current moment (state-anxiety scale). Total scores range from 20 to 80, with higher scores indicating greater maladjustment.
Change in Depression (Beck Depression Inventory-II) | Single administration at baseline, 8 weeks, 6 month and 12 follow up
  BDI contains 21 items that measure severity of depressive symptomatology on a three-point scale (0 = absence of symptoms, 3 = most severe). Respondents answer for the previous week. Total scores range from 0 to 63. Ranges for clinical levels of depression are 0 to 13 (minimal), 14 to 19 (mild), 20 to 28 (moderate), and 29 to 63 (severe).
Change in 36-Item Short Form Survey (SF-36) | Single administration at baseline, 8 weeks, 6 month and 12 follow up
  The SF-36 is a 36-item scale that assesses health status and quality of life The SF-36 includes eight domains: limitations in physical activities because of health problems; limitations in social activities because of physical or emotional problems; limitations in usual role activities because of physical health problems); bodily pain; general mental health (psychological distress and well-being); limitations in usual role activities because of emotional problems; vitality (energy and fatigue); and general health perceptions. Participants respond based on how they have felt over the previous week. The items use Likert-type scales, some with 5 or 6 points and others with 2 or 3 points. The SF-36 is a sensitive indicator of CG mental and physical health.
Change in Caregiver Burden (Zarit Burden Scale) | Single administration at baseline, 8 weeks, 6 month and 12 follow up
  Self-report measure of caregiver burden. 12-item scale that asks caregivers to rate from never (0) to nearly always (4) how often they experience feelings of stress or burden across various aspects and situations of caregiving.
Change in Cognitive Failures Questionnaire (CFQ) | Single administration at baseline, 8 weeks, 6 month and 12 follow up
  A 25-item scale measuring subjective cognition. Caregivers rate on a scale of 0 (never) to 4 (very often) how often they experience cognitive mistakes and errors in daily tasks.
Change in Dementia Patient's Caregiver Quality of Life Scale | Single administration at baseline, 8 weeks, 6 month and 12 follow up
  A 20-item questionnaire measuring the CG's quality of life.
Change in Objective Wake After Sleep Onset (Actigraph) | Daily at baseline, 8 weeks, 6 month and 12 follow up
  Wake after sleep onset via Actiwatch-2
Change in Objective Sleep Onset Latency (Actigraph) | Daily at baseline, 8 weeks, 6 month and 12 follow up
  Sleep Onset Latency via Actiwatch-2
Change in Objective Sleep Efficiently (Actigraph) | Daily at baseline, 8 weeks, 6 month and 12 follow up
  Sleep Efficiency via Actiwatch-2
Change in NIH Toolbox | Single administration at baseline, 8 weeks, 6 month and 12 follow up
  Caregivers will complete this 20-min computerized battery in single sitting. Domains tested include processing speed and attention, visuospatial ability and memory, verbal learning and memory, and executive functioning and working memory. Cognitive domains tested are ones that research has shown are impacted by caregiving.
Change in Daily Joggle Battery | Daily at baseline, 8 weeks, 6 month and 12 follow up
  Completed each morning (~15-mins) for 7 days during each assessment period. Caregivers will complete this online neuropsychological battery. Practice effects limited by: 16 versions, randomized presentation order, and 12 or more wks before repeating any version. Domains tested include processing speed and attention, visuospatial ability and memory, verbal learning and memory, and executive functioning and working memory. Cognitive domains tested are ones that research has shown are impacted by caregiving. Daily testing enhances ecological validity.

OTHER OUTCOMES:
Change in Neuropsychiatric Inventory(NPI) Nighttime Behavior Scale | Single administration at baseline, 8 weeks, 6 month and 12 follow up
  CG indicates the frequency and severity of 8 nighttime behaviors of the PWD (difficulty falling asleep, wandering during the night, etc.), as well as the level of emotional distress they experience associated with each behavior.
Change in Dementia Severity Rating Scale | Single administration at baseline, 8 weeks, 6 month and 12 follow up
  CG rates severity of dementia across several domains: memory, speech and language, recognition of family members, orientation to place and time, ability to make decisions, social and community activity, home activities and responsibilities, personal care, eating, control or urination and bowels, ability to get from place to place. Higher scores indicate more severe dementia.
Change in Patient-Caregiver Functional Unit Scale (PCFUS) | Single administration at baseline, 8 weeks, 6 month and 12 follow up
  Questionnaire that assesses the stability of the CG/PWD dyad for 14 activities of daily living and instrumental activities of daily living. CG respondents indicate the patient's functional ability, whether the CG assists with the task, and whether the CG has emotional or physical difficulty assisting with the task
Change in Godin Leisure-Time Exercise Questionnaire | Single administration at baseline, 8 weeks, 6 month and 12 follow up
  This 4-item self-administered questionnaire assesses the number of times one engages in mild, moderate and strenuous LTPA bouts of at least 15 min duration in a typical week.
Satisfaction Survey | Single administration at post-treatment - 8 weeks
  Experience with the assessments, procedures, and other features of the research study; score range: 9-90 (low satisfaction - high satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Christina S McCrae, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ory MG, Hoffman RR 3rd, Yee JL, Tennstedt S, Schulz R. Prevalence and impact of caregiving: a detailed comparison between dementia and nondementia caregivers. Gerontologist. 1999 Apr;39(2):177-85. doi: 10.1093/geront/39.2.177. PMID 10224714
- [Background] Rowe MA, McCrae CS, Campbell JM, Benito AP, Cheng J. Sleep pattern differences between older adult dementia caregivers and older adult noncaregivers using objective and subjective measures. J Clin Sleep Med. 2008 Aug 15;4(4):362-9. PMID 18763429
- [Background] Vitaliano PP, Murphy M, Young HM, Echeverria D, Borson S. Does caring for a spouse with dementia promote cognitive decline? A hypothesis and proposed mechanisms. J Am Geriatr Soc. 2011 May;59(5):900-8. doi: 10.1111/j.1532-5415.2011.03368.x. PMID 21568959
- [Background] Joling KJ, van Hout HP, Schellevis FG, van der Horst HE, Scheltens P, Knol DL, van Marwijk HW. Incidence of depression and anxiety in the spouses of patients with dementia: a naturalistic cohort study of recorded morbidity with a 6-year follow-up. Am J Geriatr Psychiatry. 2010 Feb;18(2):146-53. doi: 10.1097/JGP.0b013e3181bf9f0f. PMID 20104070
- [Background] Markowitz JS, Gutterman EM, Sadik K, Papadopoulos G. Health-related quality of life for caregivers of patients with Alzheimer disease. Alzheimer Dis Assoc Disord. 2003 Oct-Dec;17(4):209-14. doi: 10.1097/00002093-200310000-00003. PMID 14657784
- [Background] Curtis AF, Williams JM, McCoy KJM, McCrae CS. Chronic Pain, Sleep, and Cognition in Older Adults With Insomnia: A Daily Multilevel Analysis. J Clin Sleep Med. 2018 Oct 15;14(10):1765-1772. doi: 10.5664/jcsm.7392. PMID 30353817
- [Background] McCrae CS, Dzierzewski JM, McNamara JP, Vatthauer KE, Roth AJ, Rowe MA. Changes in Sleep Predict Changes in Affect in Older Caregivers of Individuals with Alzheimer's Dementia: A Multilevel Model Approach. J Gerontol B Psychol Sci Soc Sci. 2016 May;71(3):458-62. doi: 10.1093/geronb/gbu162. Epub 2014 Nov 26. PMID 25429026
- [Background] McCrae CS, Vatthauer KE, Dzierzewski JM, Marsiske M. Habitual Sleep, Reasoning, and Processing Speed in Older Adults with Sleep Complaints. Cognit Ther Res. 2012 Apr;36(2):156-164. doi: 10.1007/s10608-011-9425-4. PMID 23243328
- [Background] Livingston WS, Rusch HL, Nersesian PV, Baxter T, Mysliwiec V, Gill JM. Improved Sleep in Military Personnel is Associated with Changes in the Expression of Inflammatory Genes and Improvement in Depression Symptoms. Front Psychiatry. 2015 Apr 30;6:59. doi: 10.3389/fpsyt.2015.00059. eCollection 2015. PMID 25983695
- [Background] Heinzelmann M, Lee H, Rak H, Livingston W, Barr T, Baxter T, Scattergood-Keepper L, Mysliwiec V, Gill J. Sleep restoration is associated with reduced plasma C-reactive protein and depression symptoms in military personnel with sleep disturbance after deployment. Sleep Med. 2014 Dec;15(12):1565-70. doi: 10.1016/j.sleep.2014.08.004. Epub 2014 Sep 10. PMID 25311836
- [Derived] McCrae CS, Curtis AF, Cottle A, Beversdorf DB, Shenker J, Mooney BP, Popescu M, Rantz M, Groer M, Stein P, Golzy M, Stearns MA, Simenson A, Nair N, Rowe MA. Impact of Web-Based Cognitive Behavioral Therapy for Insomnia on Stress, Health, Mood, Cognitive, Inflammatory, and Neurodegenerative Outcomes in Rural Dementia Caregivers: Protocol for the NiteCAPP CARES and NiteCAPP SHARES Randomized Controlled Trial. JMIR Res Protoc. 2022 Jun 14;11(6):e37874. doi: 10.2196/37874. PMID 35700020